CLINICAL TRIAL: NCT06056531
Title: The Effect of First Attempts at the Success of Peripheral Intravenous Cannulation Using Three Different Techniques on Nursing Students: A Randomized Controlled Trial
Brief Title: Peripheral Intravenous Cannulation Using Three Different Techniques on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Hulya Yilmaz, Principal Investigator, PhD, Msc, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22/09/2021-13/22
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Image; Knowledge, Attitudes, Practice
Keywords: peripheral intravenous cannulation; infrared light; isometric exercise
MeSH Terms: conditions — Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized controlled experimental study.
Masking Description: Because of the nature of the device and the procedure of venipuncture, blinding could not be performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIR light visualization (Experimental): The participant performing PVC carried out the procedure on the arm vein of another volunteer classmate with the help of vein imaging by NIR. All interventions were conducted under the observation of the researchers. The researchers used a chronometer to measure and record how long the PVC took. Participants were asked about the degree of vein prominence under NIR light after the tourniquet was applied, using inspection and palpation. The chronometer was started after the tourniquet was applied and stopped when the catheter plaster was applied. The time that it took to choose the materials needed for the PVC was not added to this time. The researchers recorded whether the PVC procedure was successful or unsuccessful. The cannula's placement during PVC was evaluated by drawing blood and returning it to the vein with a syringe. The PVC procedure was considered a failure if the vein was not opened or no blood reached the syringe.
  Interventions: Other: Near infrared light imaging
- isometric hand exercise (Experimental): In this group, the participants performing PVC carried out the procedure by observing vein dilation after isometric exercise. Before the procedure, the students on whom PVC was to be performed were given two stress balls, and they were told how to use them for 15 minutes. The stress balls used in the study were 6 cm in diameter and yellow in color. They were of medium hardness and made of high-quality silicone. The participants were told to squeeze and relax the stress ball in the palm of their hands after counting from one to three, to continue doing this until the procedure began, and to concentrate on squeezing the ball. Participants were asked about the degree of vein prominence after the isometric exercise and tourniquet was applied, using inspection and palpation. The remaining stages were carried out in the same way as with all of the groups.
  Interventions: Other: Isometric exercise with stress ball
- Control group: no intervention (No Intervention): The students in this group performed the PVC procedure directly on each other's arm veins without NIR or isometric exercise. Participants were asked about the degree of vein prominence after the tourniquet was applied, using inspection and palpation. The remaining stages were carried out in the same way as with all of the groups.

INTERVENTIONS:
Other: Near infrared light imaging — The participant performing PVC carried out the procedure on the arm vein of another volunteer classmate with the help of vein imaging by NIR. All interventions were conducted under the observation of the researchers.
  Arms: NIR light visualization
Other: Isometric exercise with stress ball — Before the procedure, the students on whom PVC was to be performed were given two stress balls, and they were told how to use them for 15 minutes. The participants were told to squeeze and relax the stress ball in the palm of their hands after counting from one to three, to continue doing this until the procedure began, and to concentrate on squeezing the ball.
  Arms: isometric hand exercise

SUMMARY:
Aim: The primary objective was to assess the effect of three different teaching techniques on the success of first-time peripheral intravenous cannulation (PVC) insertion as well as the vein prominence of nursing students. As a secondary objective, the authors conducted research on the students' PVC knowledge levels and skills performance, in the PVC procedure and the duration of the procedure, their satisfaction, and self-confidence in learning.

Design: A randomized controlled trial with a pretest and posttest was conducted between February and July 2022, with near-infrared light visualization (n=49), isometric exercise (n=50), and each other's arms (n=48) with nursing students in Turkey.

DETAILED DESCRIPTION:
Aim: The primary objective was to assess the effect of three different teaching techniques on the success of first-time peripheral intravenous cannulation (PVC) insertion as well as the vein prominence of nursing students. As a secondary objective, the authors conducted research on the students' PVC knowledge levels and skills performance, in the PVC procedure and the duration of the procedure, their satisfaction, and self-confidence in learning.

Methods: A randomized controlled trial with a pretest and posttest was conducted between February and July 2022, with near-infrared light visualization (n=49), isometric exercise (n=50), and each other's arms (n=48) with nursing students in Turkey.

Performing the application on the NIR light visualization group: The participants in this group were taught to use the device, previously. The NIR light device was held by the researchers at 20cm. The participant performing PVC carried out the procedure on the arm vein of another volunteer classmate with the help of vein imaging by NIR. All interventions were conducted under the observation of the researchers. Two researchers made assessments independent of each other based on the C-PVC. The researchers used a chronometer to measure and record how long the PVC took. Participants were asked about the degree of vein prominence under NIR light after the tourniquet was applied, using inspection and palpation. The chronometer was started after the tourniquet was applied and stopped when the catheter plaster was applied. The time that it took to choose the materials needed for the PVC was not added to this time. The researchers recorded whether the PVC procedure was successful or unsuccessful. The cannula's placement during PVC was evaluated by drawing blood and returning it to the vein with a syringe. The PVC procedure was considered a failure if the vein was not opened or no blood reached the syringe. The catheter was taken out, a cotton tampon was applied, and the arm was elevated for five minutes whether the PVC attempt was successful or not. The SCLS was completed immediately after the procedure.

Performing the application on the isometric exercise group: In this group, the participants performing PVC carried out the procedure by observing vein dilation after isometric exercise. Before the procedure, the students on whom PVC was to be performed were given two stress balls, and they were told how to use them for 15 minutes. The stress balls used in the study were 6 cm in diameter and yellow. They were of medium hardness and made of high-quality silicone. The participants were told to squeeze and relax the stress ball in the palm of their hands after counting from one to three, to continue doing this until the procedure began, and to concentrate on squeezing the ball. Participants were asked about the degree of vein prominence after the isometric exercise and tourniquet was applied, using inspection and palpation. The remaining stages were carried out in the same way as with all of the groups.

Control group: The students in this group performed the PVC procedure directly on each other's arm veins without NIR or isometric exercise. Participants were asked about the degree of vein prominence after the tourniquet was applied, using inspection and palpation. The remaining stages were carried out in the same way as with all of the groups.

ELIGIBILITY:
Inclusion Criteria:

* participants who did not use alcohol
* participants who did not drug abuse
* participants who completed the immunization /vaccination schedule.
* participants who volunteered to participated in the study

Exclusion Criteria:

* participants who were diagnosed with a chronic illness,
* participants who have a disorder causing bleeding,
* participants who have a psychiatric illness,
* participants who had not received vaccinations for HBV, HCV, or HIV vaccine
* participants who were pregnant
* participants who did not volunteer to participate in the study were not included in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Prominence of the selected vein (image) | 6 months
  Prominence of the vein: 1st degree : veins not visible or palpable, 2nd degree : veins visible but not palpable, 3rd degree : veins barely visible and palpable, 4th degree : veins visible and palpable, 5th degree : veins clearly visible and easily palpable.
Knowledge, attitude, practice | 6 months
  A higher total test score was interpreted as a higher level of PVC knowledge. According to the test score, which was between 0 and 40 points, a higher total test score in the assessment demonstrated that the student's PVC skills level was high.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Health Sciences Faculty of the Nursing Department, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clerkin R, Patton D, Moore Z, Nugent L, Avsar P, O'Connor T. What is the impact of video as a teaching method on achieving psychomotor skills in nursing? A systematic review and meta-analysis. Nurse Educ Today. 2022 Apr;111:105280. doi: 10.1016/j.nedt.2022.105280. Epub 2022 Jan 24. PMID 35139443
- [Result] Fukuroku K, Narita Y, Taneda Y, Kobayashi S, Gayle AA. Does infrared visualization improve selection of venipuncture sites for indwelling needle at the forearm in second-year nursing students? Nurse Educ Pract. 2016 May;18:1-9. doi: 10.1016/j.nepr.2016.02.005. Epub 2016 Feb 18. PMID 27235559
- [Result] Helm RE, Klausner JD, Klemperer JD, Flint LM, Huang E. Accepted but unacceptable: peripheral IV catheter failure. J Infus Nurs. 2015 May-Jun;38(3):189-203. doi: 10.1097/NAN.0000000000000100. PMID 25871866
- [Result] Filipovich SJ, Dilgard JW, Conrad SP, Moore CB, Hefley JB. Training Program for Ultrasound-Guided Intravenous Catheter Insertion. Mil Med. 2021 Aug 28;186(9-10):e879-e883. doi: 10.1093/milmed/usab176. PMID 33939820
- [Derived] Yilmaz H, Yilmaz D, Cinar HG. The effect of three different techniques used to improve vein prominence on the first peripheral venous catheterization experience in nursing students: a randomized controlled study. BMC Med Educ. 2025 May 22;25(1):757. doi: 10.1186/s12909-025-07350-0. PMID 40405183